CLINICAL TRIAL: NCT03330938
Title: Randomized Controlled Trial to Evaluate the Effect of a Cognitive Behavioral Program and Resilient Model in the Treatment of Depression and Anxiety and Impact on the Quality of Life in End-Stage Renal Disease Patients
Brief Title: Decreasing Depression and Anxiety and Their Effect on QoL of ESRD Patients (End-Stage Renal Disease)
Acronym: ESRD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Collaborators: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Cristina Jazmin Gonzalez Flores, Principal Investigator, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: p3wkkbgz
Record Dates: First submitted 2017-08-02; First posted 2017-11-06 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: End-Stage Renal Disease
Keywords: Hemodialysis; Resilience; Cognitive Behavioral Therapy
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, randomized clinical trial
Who Masked: Investigator
Masking Description: Evaluation measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBI and Resilience (Experimental): 8 sessions total, once a week, 2 hours long each, consistent of 6 sessions of Cognitive-behavioral Intervention (CBI) plus 2 sessions to improve resilience strengths.
  Interventions: Behavioral: CBI and Resilience
- Cognitive-behavioral Intervention (Active Comparator): 8 sessions total, once a week, 2 hours long each. Cognitive-behavioral Intervention (CBI) without resilience strengthening.
  Interventions: Behavioral: Cognitive-behavioral Intervention

INTERVENTIONS:
Behavioral: CBI and Resilience — A combination of CBI techniques (Behavioural activation with positive reinforcement, Deep breathing and muscle relaxation, Cognitive restructuring) + Resilience strengthening (Identifying resilient strengths and potentialities, plus Imagination and projection into the future).
  Arms: CBI and Resilience
Behavioral: Cognitive-behavioral Intervention — Only CBI techniques (Behavioural activation with positive reinforcement, Deep breathing and muscle relaxation, Cognitive restructuring).
  Other Names: CBI
  Arms: Cognitive-behavioral Intervention

SUMMARY:
This study evaluates the effect of a single cognitive-behavioral intervention (CBI) in a control group against the same CBI plus the strengthening of resiliency skills in an experimental group, on ESRD patients.

DETAILED DESCRIPTION:
Cognitive behavioral therapy has long been an alternative in the treatment of symptoms of depression and anxiety in patients with chronic diseases such as renal failure, however the combination of therapeutic approaches that include not only pathological but also another more positive approach (as the resilient model), represents a novel proposal for the treatment of negative psychological symptoms and improvement of the quality of life in these patients.

The inclusion of the resilient model in a cognitive behavioral intervention serves as a possibility of therapeutic target that could enhance the effectiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18, and younger than 61 years old
* Depression score in the Beck Depression Inventory (BDI) greater than 30 points.
* Anxiety score in the Beck Anxiety Inventory (BAI) greater than 40 points.
* Have not been hospitalized over the last 6 months
* Signing of informed consent

Exclusion Criteria:

* May not be able to communicate in the Spanish language.
* Presence of psychiatric comorbidity (suicide ideation or depressive or anxious).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-10-23 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Perception (change is being assessed from baseline depression, at 8 weeks and after 5 weeks). | From Baseline, at 8 weeks for the intervention phase, and 5 weeks of following.
  Outcome measuring will be held at the baseline, after finishing the intervention (8 weeks), and after a following period of 5 weeks.
  Tool: Kidney Disease Quality of life (KDQOL 36)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Martha Meda, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Cristina Jazmín Gonzalez Flores, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chan L, Tummalapalli SL, Ferrandino R, Poojary P, Saha A, Chauhan K, Nadkarni GN. The Effect of Depression in Chronic Hemodialysis Patients on Inpatient Hospitalization Outcomes. Blood Purif. 2017;43(1-3):226-234. doi: 10.1159/000452750. Epub 2017 Jan 24. PMID 28114133
- [Background] Chan R, Dear BF, Titov N, Chow J, Suranyi M. Examining internet-delivered cognitive behaviour therapy for patients with chronic kidney disease on haemodialysis: A feasibility open trial. J Psychosom Res. 2016 Oct;89:78-84. doi: 10.1016/j.jpsychores.2016.08.012. Epub 2016 Aug 29. PMID 27663114
- [Background] Duarte PS, Miyazaki MC, Blay SL, Sesso R. Cognitive-behavioral group therapy is an effective treatment for major depression in hemodialysis patients. Kidney Int. 2009 Aug;76(4):414-21. doi: 10.1038/ki.2009.156. Epub 2009 May 20. PMID 19455196
- [Background] Wang JL, Zhang DJ, Zimmerman MA. RESILIENCE THEORY AND ITS IMPLICATIONS FOR CHINESE ADOLESCENTS. Psychol Rep. 2015 Oct;117(2):354-75. doi: 10.2466/16.17.PR0.117c21z8. Epub 2015 Oct 7. PMID 26444835
- [Background] John MM, Gupta A, Sharma RK, Kaul A. Impact of residual renal function on clinical outcome and quality of life in patients on peritoneal dialysis. Saudi J Kidney Dis Transpl. 2017 Jan-Feb;28(1):30-35. doi: 10.4103/1319-2442.198109. PMID 28098100
- [Background] Lerma A, Perez-Grovas H, Bermudez L, Peralta-Pedrero ML, Robles-Garcia R, Lerma C. Brief cognitive behavioural intervention for depression and anxiety symptoms improves quality of life in chronic haemodialysis patients. Psychol Psychother. 2017 Mar;90(1):105-123. doi: 10.1111/papt.12098. Epub 2016 Jul 20. PMID 27435635
- [Background] Matzka M, Mayer H, Kock-Hodi S, Moses-Passini C, Dubey C, Jahn P, Schneeweiss S, Eicher M. Relationship between Resilience, Psychological Distress and Physical Activity in Cancer Patients: A Cross-Sectional Observation Study. PLoS One. 2016 Apr 28;11(4):e0154496. doi: 10.1371/journal.pone.0154496. eCollection 2016. PMID 27124466
- [Background] Zalai D, Szeifert L, Novak M. Psychological distress and depression in patients with chronic kidney disease. Semin Dial. 2012 Jul;25(4):428-38. doi: 10.1111/j.1525-139X.2012.01100.x. PMID 22809005